CLINICAL TRIAL: NCT00195884
Title: Resistance Exercise as an Intervention in Type 2 Diabetes Mellitus
Brief Title: Diabetes Aerobic and Resistance Exercise (DARE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Ottawa (Other); Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MCT-44155
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus
Keywords: Diabetes Mellitus; Type 2 Diabetes; Aerobic; Resistance; weight training; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aerobic Group (Experimental): Aerobic training is divided into three stages: the Starter phase (during the run-in period), the Progression phase, and the Maintenance phase. All aerobic activities are performed on a cycle ergometer, treadmill, elliptical exercise machine or stairclimber. Subjects are free to vary the machine(s) used from one visit to the next. Exercise intensity is standardized using Polar Heartminder heart rate monitors that display the subject's heart rate and emits a warming signal when heart rate is outside the prescribed training zone, thus guiding the subject in adjustment of the work load up or down to achieve the desired intensity.
  Interventions: Behavioral: Aerobic and Resistance Exercise
- Resistance Group (Experimental): Exercises are performed at weight machines arranged in a circuit. Throughout the resistance training program, subjects will alternate between the exercises of group A and group B below.
  * Group A: abdominal crunches, seated row (back), seated biceps curls, supine bench press (chest), leg press, shoulder press (shoulders and neck); leg extension (quadriceps)
  * Group B: abdominal crunches, lat pulldown (back), sitting chest press (chest), leg press, upright row (shoulders and neck), triceps pushdown, leg curls (hamstrings).
  Subjects are instructed to exhale while lifting a weight and inhale while lowering it, in order to minimize blood pressure excursions. Warm-up and cooldown are the same as for aerobic training.
  Interventions: Behavioral: Aerobic and Resistance Exercise
- Combined Aerobic and Resistance Training (Experimental): Combined aerobic and resistance training. This group will perform both aerobic and resistance training programs, as described above. The aerobic and resistance components are performed on the same days, in varying orders.
  Interventions: Behavioral: Aerobic and Resistance Exercise
- Control Group (No Intervention): Members of this group are asked to revert to their pre-study activity levels for 5 months, at which point they begin the combined aerobic and resistance exercise program.

INTERVENTIONS:
Behavioral: Aerobic and Resistance Exercise — Aerobic activities are performed on a cycle ergometer or treadmill. Exercise intensity is standardized using Polar Heart rate monitors that display the subject's heart rate.
  Resistance training:Exercises are performed at weight machines arranged in a circuit. Throughout the resistance training program, subjects will alternate between the exercises of group A and group B below.
  Group A: abdominal crunches, seated row, seated biceps curls, supine bench press, leg press, shoulder press; leg extension Group B: abdominal crunches, lat pulldown, sitting chest press, leg press, upright row, triceps pushdown, leg curls.
  Combined aerobic and resistance training group will perform both aerobic and resistance training programs, as described above.
  Control: members of this group are asked to revert to their pre-study activity levels for 5 months, at which point they begin the combined aerobic and resistance exercise program.
  Other Names: non applicable
  Arms: Aerobic Group; Combined Aerobic and Resistance Training; Resistance Group

SUMMARY:
The main purpose of this study is to assess the impact of exercise training (aerobic exercise, resistance exercise, combined aerobic and resistance exercise) versus a sedentary waiting list control on glycemic control (as reflected in reduced hemoglobin A1c [HbA1c]), body composition (weight, body mass index [BMI], waist circumference, total body fat, visceral and subcutaneous abdominal fat, mid-thigh muscle cross-sectional area), lipids (Apo-B, Apo-A1, Apo-B/A1 ratio, low density lipoprotein (LDL) particle diameter, high-sensitivity C-reactive protein) and quality of life.

DETAILED DESCRIPTION:
Background. The incidence of type 2 diabetes mellitus in the Western world is rising rapidly due to increases in obesity and sedentary behaviour, and diabetes is among the most potent common risk factors for premature disability and mortality. Landmark clinical trials such as the UK Prospective Diabetes Study proved that these excess risks in type 2 diabetes can be reduced through relatively modest improvements in glycemic control (HbA1c difference of 0.9% over time). The excess morbidity and mortality in diabetes is attributable both to hyperglycemia and to a cluster of other metabolic disturbances associated with insulin resistance, and exercise can have beneficial effects on all of these abnormalities. The standard recommendation to people with diabetes has been to perform aerobic exercise such as brisk walking, swimming, or jogging. There is very little research on resistance exercise (such as weight lifting or exercise with weight machines) in type 2 diabetes. Resistance exercise in non-diabetic subjects increases lean body mass, resulting in increased metabolic rate, decreased insulin resistance and increased glucose disposal. Furthermore, in a recent randomized trial the addition of resistance exercise to a cardiac rehabilitation program resulted in marked improvements in quality of life, to a far greater extent than seen with aerobic exercise alone. For these reasons, we feel that resistance exercise in type 2 diabetes is a modality worthy of further research. A pilot study of our present proposal, funded by the Canadian Diabetes Association (CDA) is in progress; compliance has been excellent with >90% attendance.

Primary research question: In patients with type 2 diabetes, does a 6-month resistance or aerobic training program result in improved glycemic control as reflected in reduced hemoglobin A1c (HbA1c)? Is the effect of one type of exercise additive to that of the other?

Secondary research questions: In patients with type 2 diabetes, what are the effects of each exercise modality on:

1. Body composition (assessed using gold-standard methods including CT scan and deuterium oxide), resting energy expenditure (using indirect calorimetry) and insulin resistance? To what extent do changes in these parameters mediate changes in HbA1c?
2. Important nontraditional metabolic CHD risk factors (LDL particle diameter, plasma insulin, apoprotein B, c-reactive protein, free fatty acids) and traditional metabolic CHD risk factors (HDL-C, LDL-C, triglycerides, total/HDL cholesterol ratio, BP)?
3. Health-related quality of life (QOL) as measured by the Well-Being questionnaire or the SF-36? Does modality of exercise or change in quality of life from baseline to 6 months predict frequency of exercise during the 6 months following the intervention?

Study design: Randomized controlled trial. After a 4-week supervised low-intensity exercise run-in period to test compliance, previously inactive Type 2 diabetic subjects not currently engaging in regular exercise are randomized to 4 arms: aerobic exercise 3X per week, resistance exercise 3X per week, both combined or waiting-list control. The exercise intervention takes place at YMCA branches in metropolitan Ottawa. Exercise is closely supervised and progressive in intensity and duration. Compliance is verified through direct supervision, completion of detailed exercise logs, and central automated electronic tracking of YMCA attendance through scanning of membership cards. Primary outcomes are measured at 6 months. At the end of 6 months subjects are given a maintenance program and reexamined 6 months later to assess the durability of any benefits from the exercise program. During the 6 month intervention period diet is standardized using repeated sessions with a dietitian, and doses of medications altering glucose, lipids and BP are held constant unless change is medically urgent.

Significance: The global burden of type 2 diabetes is increasing, and complications of the illness occur primarily in those whose glycemic control is fair or poor. If appropriately selected exercise training improves glycemic control and is adopted by more patients, it is likely that the morbidity associated with type 2 diabetes will be decreased. This is particularly true if such training also improves quality of life, and more people are thus inclined to continue exercising in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus as defined by the 1998 CDA Guidelines
* Male or female
* treated with diet and/or oral agents (no insulin)
* age 40-70
* HbA1c 0.066-0.099

Exclusion Criteria:

* Participation during the previous 6 months in a regular program of exercise or aerobic sports greater than 2 times per week for at least 20 minutes per session, or in any resistance training during the previous 6 months
* Insulin therapy, or uncontrolled hyperglycemia (HbA1c>0.099). Insulin therapy is an exclusion criterion because it would render HOMA insulin sensitivity calculation invalid.
* Changes in medications for diabetes, BP or lipids in the 2 months prior to enrollment.
* Significant weight change (increase or decrease of greater than 5% of body weight during the two months before enrollment).
* Significant renal disease: serum creatinine greater than 200 mEq/l. or proteinuria >1 g/24 hours.
* Uncontrolled hypertension: BP >160 mm Hg systolic or >95 mm Hg diastolic BP in a sitting position.
* Restrictions in physical activity due to disease: intermittent claudication, severe peripheral neuropathy or active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis.
* Other illness, judged by the patient or study physician to make participation in this study inadvisable.
* Significant cognitive deficit resulting in inability to understand or comply with instructions.
* Pregnancy at the start of the study, or intention to become pregnant in the next year.
* Inability to communicate in English or French.
* Unwillingness to sign informed consent.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 1999-09; Primary Completion 2005-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c (HbA1c) | 6-months
  Measured pre and post intervention

SECONDARY OUTCOMES:
Body composition (CT scan) | 6-months
  Measured pre and post intervention
resting energy expenditure | 6-months
  Measured pre and post intervention
LDL particle diameter, insulin, CRP, FFA, HDL, LDL, Total chol./HDL ratio, triglycerides | 6-months
  Measured pre and post intervention
Blood Pressure | 6-months
  Measured pre and post intervention
quality of life (QOL) | 6-months
  Measured pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Sigal, MD MPH FRCPC, Principal Investigator — Ottawa Hospital Research Institute, Ottawa Hospital, University of Ottawa
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Sigal RJ, Kenny GP, Wasserman DH, Castaneda-Sceppa C. Physical activity/exercise and type 2 diabetes. Diabetes Care. 2004 Oct;27(10):2518-39. doi: 10.2337/diacare.27.10.2518. No abstract available. PMID 15451933
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Derived] Terada T, Boule NG, Forhan M, Prado CM, Kenny GP, Prud'homme D, Ito E, Sigal RJ. Cardiometabolic risk factors in type 2 diabetes with high fat and low muscle mass: At baseline and in response to exercise. Obesity (Silver Spring). 2017 May;25(5):881-891. doi: 10.1002/oby.21808. Epub 2017 Mar 20. PMID 28317297
- [Derived] Gavin C, Sigal RJ, Cousins M, Menard ML, Atkinson M, Khandwala F, Kenny GP, Proctor S, Ooi TC; Diabetes Aerobic and Resistance Exercise (DARE) trial investigators. Resistance exercise but not aerobic exercise lowers remnant-like lipoprotein particle cholesterol in type 2 diabetes: a randomized controlled trial. Atherosclerosis. 2010 Dec;213(2):552-7. doi: 10.1016/j.atherosclerosis.2010.08.071. Epub 2010 Sep 27. PMID 20870234
- [Derived] Reid RD, Tulloch HE, Sigal RJ, Kenny GP, Fortier M, McDonnell L, Wells GA, Boule NG, Phillips P, Coyle D. Effects of aerobic exercise, resistance exercise or both, on patient-reported health status and well-being in type 2 diabetes mellitus: a randomised trial. Diabetologia. 2010 Apr;53(4):632-40. doi: 10.1007/s00125-009-1631-1. Epub 2009 Dec 13. PMID 20012857
- [Derived] Sigal RJ, Kenny GP, Boule NG, Wells GA, Prud'homme D, Fortier M, Reid RD, Tulloch H, Coyle D, Phillips P, Jennings A, Jaffey J. Effects of aerobic training, resistance training, or both on glycemic control in type 2 diabetes: a randomized trial. Ann Intern Med. 2007 Sep 18;147(6):357-69. doi: 10.7326/0003-4819-147-6-200709180-00005. PMID 17876019